CLINICAL TRIAL: NCT04060641
Title: Association Between a Multi-Gene Panel and Renal Denervation Effectiveness in Patients With Hypertension
Acronym: GxRDxHTN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geneticure, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GCERDN01
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RDN Patients: Patients who have received renal denervation with the Medtronic SymplicitySpyral device will have DNA collected in using a buccal swab.
  Interventions: Genetic: Geneticure for RDN Genetic Panel

INTERVENTIONS:
Genetic: Geneticure for RDN Genetic Panel — This retrospective trial will include the collection of DNA using buccal swabs and the assessment of 22 genotypes for scoring to assess response to renal denervation

SUMMARY:
The purpose of this study is to assess the effectiveness of a multi-gene panel to determine which subjects are likely to respond to renal denervation therapy with Medtronic's Symplicity Spyral™ multi-electrode renal denervation system.

DETAILED DESCRIPTION:
The objective of this study is to assess if renal denervation (RDN) effectiveness using the Symplicity SpyralTM multi-electrode renal denervation system is associated with ranked genomic scoring from the Geneticure multi-gene algorithm for renal denervation. The present study will assess if subjects who have a high genetic score, based on the hypothesized importance of the organ systems involved, will have differential responsiveness to RDN in a descending order. The genetic scoring is collectively ranked in a specific order, in that:

* Subjects with a "high level of general functionality" (functionality in the sympathetic nervous system (SNS), cardiac, vascular (renin-angiotensin-aldosterone system (RAAS)), and renal system genotypes will be most responsive to RDN.
* Subjects with high number of functional genotypes of SNS, cardiac, and RAAS will be the next most responsive group.
* Subjects with functionality in genotypes of SNS and cardiac systems will demonstrate the next most responsive group.
* Subjects with functionality in the SNS genotypes will demonstrate some degree of responsiveness.
* Subjects with functionality in the renal system, but not SNS, cardiac, nor RAAS, will be the least responsive to this therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is currently or has previously been enrolled in a Medtronic clinical study utilizing the Symplicity Spyral™ multi-electrode renal denervation system.
2. Subject received Renal Denervation.
3. Subject has met the primary efficacy endpoint for the Medtronic Symplicity Spyral study and which arm they were randomized to.
4. Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* Unable to provide written, informed, consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll subjects with uncontrolled hypertension, enrolled in one of Medtronic's clinical studies utilizing the Symplicity Spyral™ multi-electrode renal denervation system, and meet the inclusion/exclusion criteria listing in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between genetic scoring and RDN effectiveness using office blood pressure | 6 months
  Change in office blood pressure (mmHg) from baseline to post- renal denervation procedure in subjects who have met the primary efficacy endpoints in the Symplicity Spyral studies (3-months for the HTN-OFF MED trial and 6-months for the HTN-ON MED trial) according to ranked genetic score values.
Correlation between genetic scoring and RDN effectiveness using ambulatory blood pressure | 6 months
  Change in ambulatory blood pressure (mmHg) from baseline to post- renal denervation procedure in subjects who have met the primary efficacy endpoints in the Symplicity Spyral studies (3-months for the HTN-OFF MED trial and 6-months for the HTN-ON MED trial) according to ranked genetic score values.

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Snyder, Principal Investigator — Geneticure, LLC
Locations (1):
- Baylor Scott and White Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No